CLINICAL TRIAL: NCT04372992
Title: Multicenter Randomized Controlled Phase III Trial Comparing Ileostomy Closure Before or After Adjuvant Therapy in Patients Operated for Rectal Cancer
Brief Title: The Stoma Closure Before or After Adjuvant Therapy Trial
Acronym: STOMAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual - no restart after pandemic suspension
Sponsor: Ospedale Umberto I di Torino (Other)
Collaborators: Rete Oncologica Piemonte, Valle d'Aosta (Other)
Responsible Party: Principal Investigator, Paolo Massucco, MD, Ospedale Umberto I di Torino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ROPCR01
Record Dates: First submitted 2020-04-20; First posted 2020-05-04 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Ileostomy; Rectal Cancer
Keywords: Chemotherapy, Adjuvant; Early closure; Late closure
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicenter controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early stoma closure (Experimental): Ileostomy closure between 30 and 40 day after rectal resection
  Interventions: Other: Timing of stoma closure
- Delayed stoma closure (Active Comparator): Ileostomy closure 15 days from the end of adjuvant therapy (up to 60 days)
  Interventions: Other: Timing of stoma closure

INTERVENTIONS:
Other: Timing of stoma closure — Defining the best timing of stoma closure in relation to adjuvant therapy compliance

SUMMARY:
This is an open-label multicenter controlled trial, including 28 centers from the Rete Oncologica (Oncological Network) of Piemonte and Valle d'Aosta in Italy (http://www.reteoncologica.it). After a curative resection for rectal cancer and temporary ileostomy, 270 patients with indication to adjuvant chemotherapy will be randomized to early (before starting adjuvant treatment) or late (after adjuvant treatment completion) stoma closure. Primary end point will the compliance to adjuvant therapy. Secondary endpoint will include quality of life and bowel function evaluation, postoperative morbidity, chemotherapy toxicity, oncological outcomes and costs comparison.

DETAILED DESCRIPTION:
Diverting ileostomy is effective in reducing severity of anastomotic complications in rectal low anterior resections and it is therefore widely used especially after neoadjuvant chemoradiation treatment. In current clinical practice, in patients with indication to adjuvant chemotherapy, closure of ileostomy is usually performed after the end of the treatment. However, a prolonged presence of the ostomy can induce the onset of ostomy-related complications such as stoma prolapse, parastomal hernia, mechanical ileus, high flow dehydration and damage to renal function. The ostomy-related complications may require unplanned or prolonged hospitalization, thus increasing costs.

Furthermore, the presence of the stoma may affect quality of life, causing alteration of the body image and imposing changes in the daily routine and lifestyle.

Early closure of the ileostomy in patients without signs of postoperative fistula has therefore been proposed.

Outcomes of early closure (within one month from surgery) of diverting ileostomy were demonstrated to be equal to those of late closure (more than 12 weeks from surgery) in 2 randomized trials. Early closure may favor a better quality of life for patients, shortening the life-period with ileostomy, reduces health system economic expenditure and may represent the most desirable and convenient choice. It was also associated with better long term functional results in a randomized trial.

In patients with indication to adjuvant therapy, however, timing to closure of the ostomy (before the start, during or at the end of treatment) is still a matter of debate in terms of compliance to systemic treatment, quality of life and overall costs.

A recent multicenter retrospective study reported an increase in gastrointestinal toxicity in ostomy patients with a significant reduction in treatment compliance.

On the other hand, early closure of the ostomy could unmask anterior resection syndrome (LARS) before chemotherapy, with potential negative impact on the tolerability of the treatment, or reveal postoperative complications thus delaying chemotherapy treatment.

The trial will investigate which is the best strategy of dealing with temporary ileostomy in relation to adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with a curative resection for rectal cancer
* Presence of a temporary ileostomy
* Age >= 18 years
* Indication to adjuvant treatment
* Absence of anastomotic dehiscence (as proved by enema and/or endoscopy)
* Able to give written informed consent

Exclusion Criteria:

* ASA >3
* ECOG Performance Status >=2
* UICC stage IV
* Severe and non-controlled systemic, oncologic, or infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with good compliance to adjuvant therapy | Measured within 48 hours after the end of the last cycle of adjuvant therapy
  Composite outcome measure including timeliness and percentage of planned dose received.
  In each subject, treatment compliance is defined as good if both the following conditions are met:
  1. adjuvant therapy starting date within 10 weeks of rectal resection;
  2. total cumulative received dose (mg/m2) >=70% of planned. The percentage of participants with good compliance in both arms will be compared.

SECONDARY OUTCOMES:
Rate of stoma-related complications | All over the study duration (up to 12 months from randomization)
  Adverse events related to the presence of stoma and postoperative complication after stoma closure
Rate of chemotherapy side effects | Immediately after the end of every single cycle (each cycle duration varies from 5 to 14 days according to the chosen scheme)
  According to CTCAE classification
Quality of life 1 | At baseline, at the end of cycle 3 (regardless of the cycle duration, that varies from 5 to 14 day according to local investigators choice) and at 12 months from randomization
  Measured by EORTC C30
Quality of life 2 | At baseline, at the end of cycle 3 (regardless of the cycle duration, that varies from 5 to 14 day according to local investigators choice) and at 12 months from randomization
  Measured by EORTC CR29
Quality of life 3 | At baseline, at the end of cycle 3 (regardless of the cycle duration, that varies from 5 to 14 day according to local investigators choice) and at 12 months from randomization
  Measured by EQ-5D-3L
Bowel function | At 12 months from rectal resection
  Measured by LARS (Low Anterior Resection Syndrome) score
Overall survival | Ut to 3 years from inclusion of the last patient
  From randomization date to death from any cause or date of last contact
Progression free survival | Ut to 3 years from inclusion of the last patient
  From randomization date to progression diagnosis or date of last contact
Costs analysis | At 12 months from randomization
  Mean cumulative costs in euro of the postoperative phase including outpatient visits, hospital stay for stoma closure, hospital re-entry and expenditures for stoma care appliances based on life-days with the stoma. Excluded are costs related to adjuvant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Massucco, MD, Principal Investigator — OA Ordine Mauriziano - Torino, Italy
Locations (28):
- Italy (28):
  - Ospedale Mons. Galliano - Chirurgia Generale (Dott. Serventi), Acqui Terme, AL
  - Ospedale SS. Antonio e Biagio - Chirurgia Generale (Dott. Priora), Alessandria, AL
  - Ospedale S. Spirito - Chirurgia Generale (Dott. Amisano), Casale Monferrato, AL
  - Ospedale S. Giacomo - Chirurgia Generale (Dott. Di Somma), Novi Ligure, AL
  - Ospedale Cardinal Massaia - Chirurgia Generale (Dott. Sorisio), Asti, AT
  - Ospedale degli Infermi - Chirurgia Generale (Dott. Polastri), Biella, BI
  - Ospedale S. Croce e Carle - Chirurgia Generale (Dott. Borghi), Cuneo, CN
  - Ospedale Regina Montis Regalis - Chirurgia Generale (Dott. Gattolin), Mondovì, CN
  - Ospedale SS. Annunziata - Chirurgia Generale (Dott. Bertolino), Savigliano, CN
  - IRCCS - Chirurgia Colorettale (Dott. Ribero), Candiolo, TO
  - Ospedale di Ciriè - Chirurgia Generale (Dott. Personettaz), Cirié, TO
  - Ospedale Civile - Chirurgia Generale (Dott. Rosato), Ivrea, TO
  - Ospedale S. Croce - Chirurgia Generale (Dott. Cumbo), Moncalieri, TO
  - Ospedale S. Luigi - Chirurgia Universitaria (Prof. Degiuli), Orbassano, TO
  - Ospedale Agnelli - Chirurgia Generale (Dott. Muratore), Pinerolo, TO
  - Ospedale degli Infermi - Chirurgia Generale (Dott. Garino), Rivoli, TO
  - Ospedale Cottolengo - Chirurgia Generale (Dott. Bima), Torino, TO
  - Ospedale Humanitas Gradenigo - Chirurgia Generale (Dott. Leli), Torino, TO
  - Ospedale S. Biagio - Chirurgia Generale (Dott. Zonta), Domodossola, VB
  - Ospedale S. Andrea - Chirurgia Generale (Dott. Testa), Vercelli, VC
  - Ospedale S. Lazzaro - Chirurgia Generale (Dott. Calgaro), Alba
  - Ospedale Parini - Chirurgia Generale (Dott. Millo), Aosta
  - Ospedale Maggiore della Carità - Chirurgia Generale (Dott. Romito), Novara
  - Ospedale Maggiore della Carità - Chirurgia Universitaria (Prof. Gentilli), Novara
  - Ospedale Martini - Chirurgia Generale (Dott. Saracco), Torino
  - Ospedale Mauriziano - Chirurgia Generale (Dott. Ferrero), Torino
  - Ospedale Molinette - Chirurgia Generale (Dott. De Paolis), Torino
  - Ospedale Molinette - Chirurgia Universitaria (Prof. Morino), Torino

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD will be available for 36 months after the results publication upon request to the principal investigator. Data will be provided in an electronic dataset containing deidentified participant files by the Unit of Epidemiology of the Azienda Ospedaliera Universitaria Città della Salute e della Scienza, Turin (Italy) after evaluation and approval of the request by the trial steering committee.
Supporting Information: Study Protocol, SAP
Time Frame: For 36 months after trial results publication
Access Criteria: Address data sharing request to the principal investigator. All requests will be evaluated and must be approved by the trial steering committee.

REFERENCES:
- [Background] Montedori A, Cirocchi R, Farinella E, Sciannameo F, Abraha I. Covering ileo- or colostomy in anterior resection for rectal carcinoma. Cochrane Database Syst Rev. 2010 May 12;2010(5):CD006878. doi: 10.1002/14651858.CD006878.pub2. PMID 20464746
- [Background] Malik T, Lee MJ, Harikrishnan AB. The incidence of stoma related morbidity - a systematic review of randomised controlled trials. Ann R Coll Surg Engl. 2018 Sep;100(7):501-508. doi: 10.1308/rcsann.2018.0126. Epub 2018 Aug 16. PMID 30112948
- [Background] Brown H, Randle J. Living with a stoma: a review of the literature. J Clin Nurs. 2005 Jan;14(1):74-81. doi: 10.1111/j.1365-2702.2004.00945.x. PMID 15656851
- [Background] Herrle F, Sandra-Petrescu F, Weiss C, Post S, Runkel N, Kienle P. Quality of Life and Timing of Stoma Closure in Patients With Rectal Cancer Undergoing Low Anterior Resection With Diverting Stoma: A Multicenter Longitudinal Observational Study. Dis Colon Rectum. 2016 Apr;59(4):281-90. doi: 10.1097/DCR.0000000000000545. PMID 26953986
- [Background] Alves A, Panis Y, Lelong B, Dousset B, Benoist S, Vicaut E. Randomized clinical trial of early versus delayed temporary stoma closure after proctectomy. Br J Surg. 2008 Jun;95(6):693-8. doi: 10.1002/bjs.6212. PMID 18446781
- [Background] Danielsen AK, Park J, Jansen JE, Bock D, Skullman S, Wedin A, Marinez AC, Haglind E, Angenete E, Rosenberg J. Early Closure of a Temporary Ileostomy in Patients With Rectal Cancer: A Multicenter Randomized Controlled Trial. Ann Surg. 2017 Feb;265(2):284-290. doi: 10.1097/SLA.0000000000001829. PMID 27322187
- [Background] Park J, Angenete E, Bock D, Correa-Marinez A, Danielsen AK, Gehrman J, Haglind E, Jansen JE, Skullman S, Wedin A, Rosenberg J. Cost analysis in a randomized trial of early closure of a temporary ileostomy after rectal resection for cancer (EASY trial). Surg Endosc. 2020 Jan;34(1):69-76. doi: 10.1007/s00464-019-06732-y. Epub 2019 Mar 25. PMID 30911920
- [Background] Keane C, Park J, Oberg S, Wedin A, Bock D, O'Grady G, Bissett I, Rosenberg J, Angenete E. Functional outcomes from a randomized trial of early closure of temporary ileostomy after rectal excision for cancer. Br J Surg. 2019 Apr;106(5):645-652. doi: 10.1002/bjs.11092. Epub 2019 Feb 1. PMID 30706439
- [Background] Tulchinsky H, Shacham-Shmueli E, Klausner JM, Inbar M, Geva R. Should a loop ileostomy closure in rectal cancer patients be done during or after adjuvant chemotherapy? J Surg Oncol. 2014 Mar;109(3):266-9. doi: 10.1002/jso.23493. Epub 2013 Nov 19. PMID 24249401
- [Background] Robertson JP, Wells CI, Vather R, Bissett IP. Effect of Diversion Ileostomy on the Occurrence and Consequences of Chemotherapy-Induced Diarrhea. Dis Colon Rectum. 2016 Mar;59(3):194-200. doi: 10.1097/DCR.0000000000000531. PMID 26855393
- [Background] Siassi M, Hohenberger W, Losel F, Weiss M. Quality of life and patient's expectations after closure of a temporary stoma. Int J Colorectal Dis. 2008 Dec;23(12):1207-12. doi: 10.1007/s00384-008-0549-2. Epub 2008 Aug 7. PMID 18685854
- [Background] Chow A, Tilney HS, Paraskeva P, Jeyarajah S, Zacharakis E, Purkayastha S. The morbidity surrounding reversal of defunctioning ileostomies: a systematic review of 48 studies including 6,107 cases. Int J Colorectal Dis. 2009 Jun;24(6):711-23. doi: 10.1007/s00384-009-0660-z. Epub 2009 Feb 17. PMID 19221766
- [Background] Hofheinz RD, Wenz F, Post S, Matzdorff A, Laechelt S, Hartmann JT, Muller L, Link H, Moehler M, Kettner E, Fritz E, Hieber U, Lindemann HW, Grunewald M, Kremers S, Constantin C, Hipp M, Hartung G, Gencer D, Kienle P, Burkholder I, Hochhaus A. Chemoradiotherapy with capecitabine versus fluorouracil for locally advanced rectal cancer: a randomised, multicentre, non-inferiority, phase 3 trial. Lancet Oncol. 2012 Jun;13(6):579-88. doi: 10.1016/S1470-2045(12)70116-X. Epub 2012 Apr 13. PMID 22503032
- [Background] Glynne-Jones R, Counsell N, Quirke P, Mortensen N, Maraveyas A, Meadows HM, Ledermann J, Sebag-Montefiore D. Chronicle: results of a randomised phase III trial in locally advanced rectal cancer after neoadjuvant chemoradiation randomising postoperative adjuvant capecitabine plus oxaliplatin (XELOX) versus control. Ann Oncol. 2014 Jul;25(7):1356-1362. doi: 10.1093/annonc/mdu147. Epub 2014 Apr 8. PMID 24718885
- [Derived] Massucco P, Fontana A, Mineccia M, Perotti S, Ciccone G, Galassi C, Giuffrida MC, Marino D, Monsellato I, Paris MK, Perinotti R, Racca P, Monagheddu C, Saccona F, Ponte E, Mistrangelo M, Santarelli M, Tomaselli F, Reddavid R, Birolo S, Calabro M, Pipitone N, Panier Suffat L, Carrera M, Potente F, Brunetti M, Rimonda R, Adamo V, Piscioneri D, Cravero F, Serventi A, Giaminardi E, Mazza L, Bellora P, Colli F, De Rosa C, Battafarano F, Trapani R, Mellano A, Gibin E, Bellomo P. Prospective, randomised, multicentre, open-label trial, designed to evaluate the best timing of closure of the temporary ileostomy (early versus late) in patients who underwent rectal cancer resection and with indication for adjuvant chemotherapy: the STOMAD (STOMa closure before or after ADjuvant therapy) randomised controlled trial. BMJ Open. 2021 Feb 19;11(2):e044692. doi: 10.1136/bmjopen-2020-044692. PMID 33608405